CLINICAL TRIAL: NCT00934700
Title: Neuroprotective Effects of Hypothermia Combined With Inhaled Xenon Following Perinatal Asphyxia
Acronym: TOBYXe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: University College London Hospitals (Other); Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: prot-002-2009
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Results first posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Hypoxic Ischaemic Encephalopathy
Keywords: perinatal asphyxia; encephalopathy; neuroprotection
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Brain Diseases | interventions — Lasers, Gas

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- Combination of hypothermia and xenon (Experimental): Combination of hypothermia and inhaled xenon
  Interventions: Other: Xenon gas
- Hypothermia and standard intensive care (No Intervention): Hypothermia and standard intensive care

INTERVENTIONS:
Other: Xenon gas — 30% Xenon gas inhaled for 24 hours
  Other Names: LENOXe
  Arms: Combination of hypothermia and xenon

SUMMARY:
This is a randomised controlled trial in newborn infants with perinatal asphyxial encephalopathy assessing whether a combination of hypothermia and inhaled xenon preserve cerebral metabolism and structure.

DETAILED DESCRIPTION:
The study hypothesis is that: Following perinatal asphyxia treatment with a combination of hypothermia and inhaled xenon preserves cerebral metabolism and structure. Following informed parental consent, infants that continue to require endotracheal tube ventilation following resuscitation will be randomised to treatment with hypothermia only or hypothermia and xenon. All infants in both groups will be treated with hypothermia for 72 hours started within 6 hours of delivery and infants allocated to hypothermia and xenon will also receive 30% xenon (balanced with oxygen and air) for 24 hours through a purpose designed delivery system. Structured neurological examination will be done daily during the 1st week after birth and at discharge. MRS and MRI will be performed once between 4-10 days of age. MRS/MRI data analysis will be by investigators blinded to the allocated intervention.

ELIGIBILITY:
Inclusion Criteria:

Infants will be eligible for enrolment into the trial if each of the following criteria is fulfilled:

* Infants 36 to 43 weeks gestation with at least one of the following:

  * Apgar score of <5 at 10 minutes after birth;
  * Continued need for resuscitation, including endotracheal or mask ventilation, at 10 minutes after birth;
  * Acidosis defined as pH <7.00 and/or base deficit >15 mmol/L in umbilical cord blood sample or any blood sample within 60 minutes of birth (arterial or venous blood).
* Moderate to severe encephalopathy consisting of altered state of consciousness (reduced or absent response to stimulation) and hypotonia, and abnormal primitive reflexes (weak or absent suck or Moro response). Clinical severity of HIE will be assessed by Thompson encephalopathy score, and modified Sarnat score.
* At least 30 minutes duration of amplitude integrated EEG (aEEG) recording that shows moderately abnormal or suppressed background aEEG activity or seizures

Exclusion Criteria:

* If treatment with hypothermia is delayed beyond 6 hours, or infants are expected to be >12 hours of age at the time of randomisation; Infants with ventilatory oxygen requirement > 70%; Attending clinician considers infant not suitable to participate because of other serious congenital abnormalities, or the infant's condition appears terminal.

Ages: 1 Hour to 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2012-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Azzopardi, MD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Academic Healthcare Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Azzopardi D, Robertson NJ, Bainbridge A, Cady E, Charles-Edwards G, Deierl A, Fagiolo G, Franks NP, Griffiths J, Hajnal J, Juszczak E, Kapetanakis B, Linsell L, Maze M, Omar O, Strohm B, Tusor N, Edwards AD. Moderate hypothermia within 6 h of birth plus inhaled xenon versus moderate hypothermia alone after birth asphyxia (TOBY-Xe): a proof-of-concept, open-label, randomised controlled trial. Lancet Neurol. 2016 Feb;15(2):145-153. doi: 10.1016/S1474-4422(15)00347-6. Epub 2015 Dec 19. PMID 26708675
- [Derived] Shankaran S. Outcomes of hypoxic-ischemic encephalopathy in neonates treated with hypothermia. Clin Perinatol. 2014 Mar;41(1):149-59. doi: 10.1016/j.clp.2013.10.008. PMID 24524452

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination of Hypothermia and Xenon: Combination of 72 hours of whole body cooling to 33.5 rectal and 30% Xenon gas inhaled for 24 hours
- Hypothermia and Standard Intensive Care: 72 hours of whole body cooling to 33.5 rectal and standard intensive care
Period: Overall Study
Arm/Group | Combination of Hypothermia and Xenon | Hypothermia and Standard Intensive Care
Started | 46 | 46
Completed | 33 | 34
Not Completed | 13 | 12
Not completed — missing scan | 5 | 9
Not completed — Death | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Combination of Hypothermia and Xenon: Combination of whole body cooling to 33.5 rectal and 30% Xenon gas inhaled for 24 hours
- Total: Total of all reporting groups
Arm/Group | Combination of Hypothermia and Xenon | Hypothermia and Standard Intensive Care | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Continuous [Mean (Standard Deviation); unit: weeks, gestation] — Gestation at delivery in weeks
  weeks, gestation | 39.8 (1.7) | 39.8 (1.3) | 39.8 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 25 | 45
  Male | 26 | 21 | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 46 | 46 | 92

OUTCOME MEASURES:

1. Primary Outcome: Lactate (Lac) / N Acetyl Aspartate (NAA) Ratio on Magnetic Resonance Spectroscopy
Description: Cerebral Lac/NAA ratio measured by magnetic resonance spectroscopy in patents
Time Frame: 10 days
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Groups:
- Combination of Hypothermia and Xenon: Combination of whole body cooling to 33.5 rectal and hypothermia and 30% Xenon gas inhaled for 24 hours
Arm/Group | Combination of Hypothermia and Xenon | Hypothermia and Standard Intensive Care
Number analyzed (Participants) | 33 | 34
ratio | 0.25 (1.30) | 0.28 (1.45)

2. Primary Outcome: Cerebral Fractional Anisotropy Measured by Diffusion Weighted Magnetic Resonance Imaging
Description: Fractional anisotropy (FA) is a measure of tissue integrity in white matter tracts measured by diffusion tensor MRI, and it has been used in work in animals to assess potential neuroprotectants and can be used to predict subsequent neurological outcomes after birth asphyxia, including in infants treated with moderate hypothermia.
  It is a scalar value between 0-1 that describe anisotropy of a diffusion process. A value of zero means that diffusion is unrestricted (or equally restricted) in all directions. A value of one means that diffusion occurs only along one axis and is fully restricted along all other directions" or similar.
  Fractional anisotropy data were extracted froma mask of the posterior limb of the internal capsule via tract-based spatial statistics. *Coefficient of variation=√(exp(var)-1), where var is the variance on the log scale
Time Frame: 10 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combination of Hypothermia and Xenon | Hypothermia and Standard Intensive Care
Number analyzed (Participants) | 30 | 33
units on a scale | 0.40 (0.05) | 0.40 (0.05)

3. Secondary Outcome: Amiel Tison Evaluation at Hospital Discharge
Description: Amiel Tison neurological assessment at discharge from hospital. Amiel Tison evaluation was developed to detect transient and permanent abnormalities in an infant's neuromotor development. Its main focus is to examine active and passive muscle tone.
Time Frame: At discharge from hospital
Population: Infants survivors at time of hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Combination of Hypothermia and Xenon | Hypothermia and Standard Intensive Care
Number analyzed (Participants) | 35 | 37
Participants
  Normal or mildly abnormal | 30 | 29
  Moderately abnormal | 3 | 7
  Very abnormal | 2 | 1

ADVERSE EVENTS:
Time Frame: 10days
Arm/Group | Combination of Hypothermia and Xenon | Hypothermia and Standard Intensive Care
All-Cause Mortality (participants affected / at risk) | 11/46 | 9/46
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 2/46 | 0/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination of Hypothermia and Xenon (N=46) | Hypothermia and Standard Intensive Care (N=46)
Subcutaneous fat necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Transient desaturation during MRI scan (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes